CLINICAL TRIAL: NCT04011241
Title: Relative Bioavailability of a Single Oral Dose of BI 1323495 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, One-way Crossover Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 1323495 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1405-0009; 2019-001570-28 (EudraCT Number)
Record Dates: First submitted 2019-07-05; First posted 2019-07-08 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference - BI 1323495 alone (Experimental): Single oral dose of 10 milligrams (mg) of film-coated tablet of BI 1323495 was administered once on day 1 in the first treatment period (period 1, visit 2) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment R.
  Interventions: Drug: BI 1323495
- Test - BI 1323495 + Itraconazole (Experimental): Single oral dose of 200 mg itraconazole (oral solution, 20 milliliter (mL) per day with 10 mg/mL) was administered once daily with 240 mL of water after an overnight fast of 9 hours (h) from day -3 to day 7 (total: 10 doses) in the second treatment period (period 2, visit 3) together with a single oral dose of 10 mg BI 1323495 administered 1 h after itraconazole administration with 240 mL of water after an overnight fast of 10 h on the fourth day of the itraconazole treatment (day 1, period 2, visit 3) as test treatment T.
  Interventions: Drug: BI 1323495; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 1323495 — Tablet
Drug: Itraconazole — Oral solution
  Arms: Test - BI 1323495 + Itraconazole

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 1323495 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test,T) as compared to when given alone as oral single dose (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* further inclusion criteria apply

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR), or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, blood coagulation, or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Current or history of relevant kidney, urinary tract diseases or abnormalities (e.g. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure)
* Estimated glomerular filtration rate according to CKD-EPI formula < 90 mL/min at screening
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* History of drug induced liver injury
* Liver enzymes (ALT, AST, GGT) above upper limit of normal at the screening examination
* History of heart failure, or any evidence of ventricular dysfunction
* Known sorbitol/polyols intolerance
* Subjects with female partner of childbearing potential who are unwilling to use male contraception (condom or sexual abstinence) from first administration until 30 days after last administration of trial medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label, two-treatment, two-period, one-way fixed-sequence design to investigate the relative bioavailability of a single oral dose of BI 1323495 when given alone (Period 1) as reference treatment (R) or in combination with itraconazole (Period 2) as test treatment (T) in healthy male subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1323495 (R) / BI 1323495 + Itraconazole (T): A single oral dose of 10 milligrams (mg) BI 1323495, film-coated tablet, was administered once on day 1, period 1, visit 2, as reference treatment R, followed by a washout period of at least 7 days, followed by period 2, visit 3, in which a single oral dose of 200 mg itraconazole (oral solution, 20 milliliter (mL) per day with 10 mg/mL) was administered once daily from day -3 to day 7, in total 10 doses. On day 1 of visit 3, 4th day of itraconazole treatment, a single oral dose of 10 mg BI 132345 was administered 1 hour (h) after itraconazole administration as test treatment T.
  BI 1323495 and itraconazole were orally administered with 240 mL of water after an overnight fast of at least 10 h for BI 1323495 and 9 h for itraconazole.
Period: Treatment Period 1
Arm/Group | BI 1323495 (R) / BI 1323495 + Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0
Period: Washout Period
Arm/Group | BI 1323495 (R) / BI 1323495 + Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0
Period: Treatment Period 2
Arm/Group | BI 1323495 (R) / BI 1323495 + Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included participants who were entered and treated with at least 1 dose of trial drug.
Arm/Group | BI 1323495 (R) / BI 1323495 + Itraconazole (T)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz)
Time Frame: Within 3 hours (h) prior and 0.33, 0.67, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 34, 47, 71, 95 (period 1) and additional 119, 143, 167h (period 2) after administration.
Population: Pharmacokintetic parameter analysis set (PKS): Participants in the treated set (TS) with at least 1 primary or secondary pharmacokinetic (PK) endpoint who were not excluded due to a protocol deviation relevant to the evaluation of PK or PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles * hour per Liter
Groups:
- BI 1323495 (R): Single oral dose of 10 milligrams (mg) of film-coated tablet of BI 1323495 was administered once on day 1 in the first treatment period (period 1, visit 2) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment R.
- BI 1323495 + Itraconazole (T): Single oral dose of 200 mg itraconazole (oral solution, 20 milliliter (mL) per day with 10 mg/mL) was administered once daily with 240 mL of water after an overnight fast of 9 hours (h) from day -3 to day 7 (total: 10 doses) in the second treatment period (period 2, visit 3) together with a single oral dose of 10 mg BI 1323495 administered 1 h after itraconazole administration with 240 mL of water after an overnight fast of 10 h on the fourth day of the itraconazole treatment (day 1, period 2, visit 3) as test treatment T.
Arm/Group | BI 1323495 (R) | BI 1323495 + Itraconazole (T)
Number analyzed (Participants) | 14 | 14
Nanomoles * hour per Liter | 124.15 (NA) — Adjusted Geometric Standard Error = 1.29 | 215.66 (NA) — Adjusted Geometric Standard Error = 1.29
Statistical Analysis 1: Comparison: BI 1323495 (R) vs BI 1323495 + Itraconazole (T); Test type: Other — Relative bioavailability; ANOVA; The statistical model was analysis of variance (ANOVA) on the logarithmic scale considering the effects "subjects" as random and "treatment" as fixed; Ratio of the geometric means (T/R) % = 173.71, 90% CI 2-sided [154.58 to 195.21] — Intra-individual geometric coefficient of variation (gCV%) = 17.6

2. Primary Outcome: Maximum Measured Concentration of BI 1323495 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles per Liter
Arm/Group | BI 1323495 (R) | BI 1323495 + Itraconazole (T)
Number analyzed (Participants) | 14 | 14
Nanomoles per Liter | 10.49 (NA) — Adjusted Geometric Standard Error = 1.23 | 14.41 (NA) — Adjusted Geometric Standard Error = 1.23
Statistical Analysis 1: Comparison: BI 1323495 (R) vs BI 1323495 + Itraconazole (T); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 137.40, 90% CI 2-sided [120.84 to 156.24] — Intra-individual geometric coefficient of variation (gCV%) = 19.4

3. Secondary Outcome: Area Under the Concentration-time Cure of BI 1323495 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time cure of BI 1323495 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomoles * hour per Liter
Arm/Group | BI 1323495 (R) | BI 1323495 + Itraconazole (T)
Number analyzed (Participants) | 13 | 10
Nanomoles * hour per Liter | 178.29 (NA) — Adjusted Geometric Standard Error = 1.24 | 300.66 (NA) — Adjusted Geometric Standard Error = 1.25
Statistical Analysis 1: Comparison: BI 1323495 (R) vs BI 1323495 + Itraconazole (T); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 168.64, 90% CI 2-sided [145.59 to 195.34] — Intra-individual geometric coefficient of variation (gCV%) = 18.1

ADVERSE EVENTS:
Time Frame: BI 1323495 (BI): 1st BI administration (AD) up to 7 days (D) thereafter; Itraconazole (IT): 1st IT until 2nd AD of BI or last IT AD up to 9D if discontinuation prior to 2nd BI AD; BI + IT: 2nd BI AD up to 7D or last IT AD up to 9D, whichever was later.
Description: Safety analyses were based on the treated set (TS). The TS included all subjects who were entered and treated with at least 1 dose of trial drug.
Groups:
- BI 1323495: Single oral dose of 10 milligrams (mg) of film-coated tablet of BI 1323495 was administered once on day 1 in the first treatment period (period 1, visit2) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment R.
- Itraconazole: Single oral dose of 200 mg itraconazole (oral solution, 20 milliliter (mL) per day with 10 mg/mL) was administered once daily with 240 mL of water after an overnight fast of 9 hours (h) from day -3 to day -1 (total: 3 doses) in the second treatment period (period 2, visit 3) as test treatment T.
- BI 1323495 + Itraconazole: Single oral dose of 200 mg itraconazole (oral solution, 20 milliliter (mL) per day with 10 mg/mL) was administered once daily with 240 mL of water after an overnight fast of 9 hours (h) from day 1 to day 7 (total: 7 doses) in the second treatment period (period 2, visit 3) together with a single oral dose of 10 mg BI 1323495 administered 1 h after itraconazole administration with 240 mL of water after an overnight fast of 10 h on the fourth day of the itraconazole treatment (day 1, period 2, visit 3) as test treatment T.
Arm/Group | BI 1323495 | Itraconazole | BI 1323495 + Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 2/14 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1323495 (N=14) | Itraconazole (N=14) | BI 1323495 + Itraconazole (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT04011241/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04011241/SAP_001.pdf